CLINICAL TRIAL: NCT00288197
Title: An Open, Prospective, Uncontrolled, Multi-Center Study To Evaluate The Efficacy And Safety Of Voriconazole In Chinese Subjects With Proven Or Probable Serious Invasive Fungal Infections
Brief Title: A Study To Assess The Efficacy And Safety Of Voriconazole In Chinese Patients With Serious Deep Tissue Fungal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1501066
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Voriconazole

INTERVENTIONS:
Drug: voriconazole

SUMMARY:
To evaluate the efficacy and safety of voriconazole in Chinese patients with proven or probable deep tissue fungal infections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with proven or probable invasive fungal infections including subjects who have failed to respond to, or have an intolerance to other approved antifungal treatments and with approval for salvage treatment by Principal Investigator and Pfizer.

Exclusion Criteria:

* Subjects who are showing continuing improvement with other antifungal agents, including amphotericin B, itraconazole, nystatin, fluconazole, flucytosine and miconazole.
* Subjects with an invasive fungal infection caused by a fungus (such as Mucor) that is not in the antifungal spectrum of voriconazole.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with a Global Efficacy assessment of either "cured" or "improved" by Week 6 visit.

SECONDARY OUTCOMES:
Safety assessment during the study period (Adverse events observed between start of treatment and follow-up visit).
Percent of subjects with a Global Efficacy assessment of either "cured" or "improved" at the time when IV administration is completed

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- China (6):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Hangzhou
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501066&StudyName=A%20Study%20To%20Assess%20The%20Efficacy%20And%20Safety%20Of%20Voriconazole%20In%20Chinese%20Patients%20With%20Serious%20Deep%20Tissue%20Fungal%20Infections